CLINICAL TRIAL: NCT07287670
Title: A Phase 2 Randomized, Double-blind, Placebo-Controlled Study to Assess the Safety and Efficacy of MTX-474 in the Treatment of Participants With Diffuse Cutaneous Systemic Sclerosis (dcSSc)
Brief Title: EncompaSSc: Evaluation of MTX-474 in Participants With Diffuse Cutaneous Systemic Sclerosis (dcSSc)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mediar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTX-474-S201; 2025-523288-39 (EudraCT Number)
Record Dates: First submitted 2025-11-18; First posted 2025-12-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis
Keywords: MTX-474-S201; MTX-474; Diffuse Cutaneous Systemic Sclerosis; dcSSc participants; dcSSc; Adult; mRSS; EncompaSSc; monoclonal antibody; EphrinB2
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MTX-474 (Experimental): MTX-474
  Interventions: Biological: MTX-474
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MTX-474 — Dosage level: 4 mg/kg Unit dose strength: 50mg/ml MTX-474 is a human immunoglobulin G1 (IgG1) monoclonal antibody that binds the human EphrinB2 with high specificity and high affinity. MTX-474 is being developed as a therapy for patients with systemic sclerosis (SSc).
  Arms: MTX-474
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A Phase 2 Randomized, Double-blind, Placebo-Controlled Study of the Safety and Efficacy of MTX-474 in Participants with Diffuse Cutaneous Systemic Sclerosis (dcSSc)

DETAILED DESCRIPTION:
Participants with dcSSc who meet the study's inclusion and exclusion criteria will be randomly assigned in a 3:2 ratio to receive MTX-474 or a matching placebo by intravenous (IV) infusion. Concomitant use of one of the approved dcSSc therapies (immunosuppressive therapy, systemic glucocorticoids or other antifibrotic agents) is permitted under certain criteria. Participants randomized to the MTX-474 arm of the study will receive an IV infusion every 4 weeks, beginning at Day 0 and ending at Week 20. The End of Treatment Visit will occur at Week 24, and a Safety Follow-Up Visit will occur at Week 28, 8 weeks after the final infusion. mRSS assessments will occur at Screening, Baseline, and at all subsequent treatment visits up to and including Week 24. Spirometry will be performed at screening and Weeks 12. HRCT will be performed at screening and week 24. DLCO will be performed at Screening. Skin biopsies will be performed at Baseline and Week 12. Participants will have blood drawn for safety assessment and to assess Ephrin receptor levels at Screening, Baseline and every 4 weeks until Week 28. Blood will be drawn for serum PK analyses relative to the first and last doses of MTX-474.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of diffuse cutaneous systemic sclerosis, classified according to 2013 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR)
2. Participant is either:

   1. Within 2 years of their first non-Raynaud's symptom and their mRSS is >7; OR
   2. >2 and ≤5 years from their first non-Raynaud's symptom, their mRSS is between 10 and 30, they are negative for the RNA polymerase 3 autoantibody, and (1) they have never had any previous spontaneous improvement in skin thickening of ≥4 points by mRSS on exams performed by the same clinician, or (2) they were never clinically noted to have a meaningful spontaneous reduction in skin thickness if mRSS was never done; OR
   3. >5 and ≤10 years from their first non-Raynaud's symptom, their mRSS is between >15 and ≤25, they are negative for the RNA polymerase 3 autoantibody, and (1) they have never had any previous spontaneous improvement in skin thickening of ≥4 points by mRSS, or (2) were never clinically noted to have a meaningful spontaneous reduction in skin thickness if mRSS was never done.
3. Participant is ≥18 years of age at time of signing the ICF.
4. Able to understand the study and provide a signed, written ICF
5. Able to read and understand the language of the ICF and other study-related materials
6. Forced vital capacity (FVCpp) of ≥45 pp10
7. Have diffusing capacity of the lungs for carbon monoxide (DLCO) of ≥30 percent predicted at Screening
8. Willing and able to complete all protocol-required study visits and procedures
9. Participants of childbearing potential must have a negative serum pregnancy test at Screening.
10. All participants with reproductive potential must agree to use and follow medically approved, highly effective methods of contraception during treatment and until 5 half-lives or 125 days after the last dose, whichever is longer

Exclusion Criteria:

1. Concomitantly have another serious medical illness, which, in the opinion of the Investigator, would interfere with the participant's ability to complete the study
2. Participant is currently on immunosuppressive therapy, systemic glucocorticoids or other antifibrotic agents detailed as follows:

   1. Immunosuppresive agents: Cyclophosphamide (IV or oral if used in the 6 months prior to Screening), calcineurin inhibitors (if used in the 30 days prior to Screening), azathioprine (if used in the 30 days prior to Screening), Janus-kinase inhibitors (if used in the 30 days prior to Screening), rituximab (if used in the 6 months prior to Screening), tocilizumab (if used in the 60 days prior to Screening) or any other biologic Disease-Modifying Antirheumatic Drugs (DMARD, if used in the last 30 days or 3 half-lives prior to Screening, whichever is longer)
   2. Antifibrotic agents: nintedanib or pirfenidone (if used in the 30 days prior to Screening). Also, exclusionary if used within 3 months of Screening are tyrosine-kinase inhibitors with recognized anti-fibrotic activity (imatinib, nilotinib, etc.)
   3. Systemic glucocorticoids: equivalent doses of prednisone greater than 10 mg/day (≤10 mg/day allowed). Has received any pulse intramuscular (IM) or intravenous (IV) steroid within 1 month of Screening
   4. Other agents:

   i. mycophenolate mofetil unless on a stable dose for at least 6 months prior to Screening and there are no plans to adjust the dose during the study; ii. mycophenolic acid unless on a stable dose for at least 6 months prior to Screening and there are no plans to adjust the dose during the study; iii. hydroxychloroquine unless on a stable dose for at least 3 months prior to Screening and there are no plans to adjust the dose during the study; and iv. methotrexate unless on a stable dose for at least 3 months prior to Screening and there are no plans to adjust the dose during the study.
3. Previous or planned hematopoietic stem cell or solid organ transplantation
4. Previous treatment with chimeric antigen receptor (CAR)-T/CAR-NK therapy
5. Clinically significant PAH as determined by the Investigator at, or prior to first day of dosing (Baseline)
6. Current use of PAH medication (endothelin receptor antagonists, prostacyclin analogues, soluble guanylate cyclase stimulators) excluding calcium channel blockers and phosphodiesterase-5 inhibitors
7. Pregnant or currently breastfeeding
8. Aspartate transaminase (AST) or alanine transaminase (ALT) >2.0 upper limit of normal
9. Creatinine clearance <45mL/min
10. History of myocardial infarction, angina or congestive heart failure
11. International normalized ratio >2 or partial thromboplastin time >1.5 × upper limit of normal
12. Active infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
13. History of clinically significant thrombotic event within 12 months prior to Screening
14. Positive anticentromere antibody
15. Systemic sclerosis renal crisis within 12 months prior to Screening
16. Confirmed diagnosis of overlap syndrome, systemic lupus erythematosus with anti-double strand (ds)DNA antibody, rheumatoid arthritis with anti-cyclic citrullinated peptide (anti-CCP) antibody, or systemic sclerosis mimics (eosinophilic fasciitis, scleromyxedema) at the time of inclusion in the study
17. Known malignancy or history of malignancy within 5 years of Screening other than non-melanoma skin cancer and in situ cervical cancer
18. Major surgery within 8 weeks prior to Screening or planned surgery during study period
19. Unable to routinely access veins for blood draws and IV infusions
20. Currently receiving another experimental agent or participating in another clinical trial. If a participant has recently received another experimental agent, then the last dose must have been at least 5 half-lives or 30 days (whichever is longer) prior to Screening
21. History of myocardial infarction, angina or congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Modified Rodnan Skin Score (mRSS) | Baseline to week 24
  Mean change from baseline to week 24 in the modified Rodnan Skin Score, a clinician-assessed measure of skin thickness across 17 body areas.
  Unit of measure: Score (range 0-51)

SECONDARY OUTCOMES:
Proportion of participants with a gene signature response in skin biopsy | 12 weeks
  Proportion of participants in each arm (MTX-474 and placebo) demonstrating a dcSSc gene expression signature response on skin biopsy at Week 12.
  Unit of Measure: Participants (%)
Number of participants with clinically significant findings on physical examination, vital signs, and clinical laboratory tests | Baseline through end of study (week 28)
  Number of participants with clinically significant findings on physical examination, vital signs, and clinical laboratory tests Unit of Measure: Participants (%)
Number of participants with dose interruptions or treatment discontinuations due to adverse events | Baseline through end of study (week 28)
  Number of participants with dose interruptions or treatment discontinuations due to adverse events Unit of Measure: Participants (%)
Safety and tolerability of MTX-474 in participants with dcSSc: Number of participants with treatment-emergent adverse events (TEAEs) and treatment-related adverse events (TRAEs) | Baseline through end of study (week 28)
  Incidence, seriousness, and severity of TEAEs and TRAEs as determined by investigator assessment.
  Unit of measure: Participants (%)
Serum concentration of MTX-474 at sparse PK time points | Baseline to week 28
  Serum MTX-474 concentrations collected at predefined sparse PK time points to support population pharmacokinetic (popPK) analysis Unit of Measure: ng/mL
Clearance (CL) of MTX-474 | Baseline to week 28
  Clearance of MTX-474 calculated from serial PK sampling using noncompartmental analysis Unit of Measure: L/hour
Terminal elimination half-life (t½) of MTX-474 | Baseline to week 28
  Terminal elimination half-life of MTX-474 derived from serial PK sampling. Unit of Measure: Hours
Area under the plasma concentration-time curve (AUC) of MTX-474 | Baseline to week 28
  AUC of MTX-474 calculated from serial PK sampling using noncompartmental analysis.
  Unit of Measure: ng·h/mL

OTHER OUTCOMES:
Proportion of participants with a response on the revised American College of Rheumatology Composite Response Index in Systemic Sclerosis (rACR-CRISS) | Baseline to week 24
  Proportion of participants achieving rACR-CRISS composite response Unit of Measure: Participants (%)
Change from baseline in Physician Global Assessment (PhGA) of disease status | Baseline to week 24
  Mean change from baseline to week 24 in the physician global assessment (phGA) of disease status in each arm Unit of Measure: Units on 0-10 visual analog scale (higher score = worse disease)
Change from baseline in Patient Global Assessment (PtGA) of disease status | Baseline to week 24
  Mean change from baseline to week 24 in the patient global assessment (PtGA) of disease status in each arm Unit of Measure: Units on 0-10 visual analog scale (higher score = worse disease)
Change from baseline in percent predicted forced vital capacity (FVCpp) | Baseline to week 24
  Mean change from baseline to week 24 on percent predicted forced vital capacity (FVCpp) Unit of Measure: Percent predicted (%)
Change from baseline in quantitative interstitial lung disease (QILD) score by high-resolution computed tomography (HRCT) | Baseline to week 24
  Mean change from baseline to week 24 in the QILD score by high resolution computed tomography scan (HRCT) in each arm Unit of Measure: Units on QILD score (0-100 scale; higher score = greater fibrosis)
Change from Baseline in free EphrinB2 levels | Baseline to week 24
  Median change from baseline to Week 24 in serum free EphrinB2 levels in each treatment arm.
  Unit of Measure: pg/mL
Change from baseline in forced vital capacity (FVC) by EphrinB2 levels | Baseline to week 24
  Mean change from baseline to Week 24 in FVC, analyzed by baseline EphrinB2 levels, in the subset of participants with interstitial lung disease (ILD).
  Unit of Measure: Percent predicted (%)
Proportion of participants achieving rACR-CRISS response by EphrinB2 levels | Up to 24 weeks
  Proportion of participants achieving a response on the revised ACR Composite Response Index in Systemic Sclerosis (rACR-CRISS), stratified by baseline EphrinB2 levels.
  Unit of Measure: Participants (%)
To assess the presence, titer and impact of antidrug antibodies (ADA) against MTX-474 | Baseline to week 28
  Samples will be collected from baseline until Week 28 to assess the rate at which antibodies develop to the study drug Unit of Measure: Titer units
Change from baseline in expression of total and phosphorylated EphB2, EphB3, and EphB4 receptors in skin | Baseline to Week 12
  Mean change from baseline to Week 12 in total and phosphorylated EphB2, EphB3, and EphB4 receptor expression in skin biopsy samples.
  Unit of Measure: Relative expression units (fold change from baseline)
Change from baseline in transcriptomic profile | Baseline to Week 12
  Change from baseline to Week 12 in global transcriptomic profile via bulk RNA sequencing analysis of skin biopsies in each arm.
  Unit of Measure: Differential gene expression (log₂ fold change)
Change from baseline in serum biomarkers of organ involvement | Baseline to weeks 12 and 24
  Change from baseline to Weeks 12 and 24 in serum levels biomarkers, including but not limited to, ProC3 and IL-6 associated with organ involvement Unit of Measure: ng/mL (or unit per biomarker)
Change from baseline in fatigue symptoms (FACIT-Fatigue score) | Baseline to week 24
  Mean change from baseline to Week 24 in fatigue symptoms as measured by the Functional Assessment of Chronic Illness Therapy-Fatigue Scale.
  Unit of Measure: Units on FACIT-Fatigue scale (range 0-52; higher score = less fatigue)
Change from baseline in gastrointestinal (GI) symptoms (UCLA SCTC GIT 2.0 score) | Baseline to week 24
  Mean change from baseline to Week 24 in GI symptom burden assessed by the UCLA SCTC GIT 2.0 questionnaire.
  Unit of Measure: Units on UCLA SCTC GIT 2.0 total score (range 0-3; higher score = worse symptoms)
Change from baseline in anxiety and depression symptoms (HADS) | Baseline to week 24
  Mean change from baseline to Week 24 in symptoms of anxiety and depression measured by the HADS instrument.
  Unit of Measure: Units on Hospital Anxiety and Depression Scale (HADS total and subscale scores; range 0-21 per subscale; higher score = worse symptoms)
Change from baseline in HAQ-DI | Baseline to week 24
  Mean change from Baseline in functional disability as assessed by HAQ-DI. Unit of measure: Score (0-3 scale)

CONTACTS AND LOCATIONS:
Locations (1):
- EncompaSSc site in Newport Beach, CA 92663, Newport Beach, California, United States

IPD SHARING:
Plan to Share IPD: No